CLINICAL TRIAL: NCT04977310
Title: Prospective, Randomized-controlled, Non-blinded, Multi-center, Pilot Trial to Compare Standard-of-care LVAD Unloading Plus Heart Failure Medications Reverse-modeling Management Versus Hemodynamics-guided LVAD Unloading with the Use of the Wireless Monitoring System CardioMEMS Plus Heart Failure Medications Reverse-remodeling Management
Brief Title: TARGET-LOAD Pilot Study Comparing Hemodynamics-guided LVAD Unloading Vs. Standard of Care
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Did not receive funding from sponsor
Sponsor: STAVROS G DRAKOS (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor-Investigator, STAVROS G DRAKOS, Professor, Cardiovascular Medicine, University of Utah
Organization: University of Utah (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB_00143654
Record Dates: First submitted 2021-07-15; First posted 2021-07-26 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-11

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control (No Intervention): After LVAD implantation, patients undergo cardiac rehab and pump speed will be optimized to maximize left ventricular unloading using echocardiographic imaging and other standard-of-care practices. During the Unloading phase, patients are serially evaluated with echocardiograms to assess for cardiac recovery, and LVAD explantation performed when predefined criteria are met. After explantation, patients undergo cardiac rehab and regular follow up.
- Intervention (Experimental): After LVAD and wireless monitoring system (CardioMEMS) implantation, patients undergo cardiac rehab and pump speed will be optimized to maximize left ventricular unloading using CardioMEMS. During the Unloading phase, invasive hemodynamic guidance (via CardioMEMS) will be utilized to optimize pressure and volume unloading along with serial echocardiographic evaluations to assess for cardiac recovery, and LVAD explantation will be considered. After explantation, patients will undergo cardiac rehab and regular follow up with adjustments of HF medications based on the CardioMEMS-guided hemodynamic assessment.
  Interventions: Device: CardioMEMS

INTERVENTIONS:
Device: CardioMEMS — Cardio-MEMS-guided Post-LVAD cardiac unloading and recovery
  Arms: Intervention

SUMMARY:
This study is a prospective, randomized-controlled, non-blinded, multi-center, pilot trial to compare standard-of-care left ventricular assist device (LVAD) unloading plus heart failure (HF) medications reverse-remodeling management versus hemodynamics-guided LVAD unloading with use of the wireless monitoring system CardioMEMS plus HF medications reverse-remodeling management.

DETAILED DESCRIPTION:
LVADs are being increasingly used in end-stage heart failure patients as a bridge to transplant (BTT) or as a destination therapy (DT). Although LVAD recipients are considered to be optimally unloaded with speed optimizations following LVAD implantation, re-hospitalizations due to HF recurrence are far from negligible. Recent studies have reported that at least 35% of hospital readmissions post-LVAD implantation are due to HF exacerbations, volume status changes or other cardiac causes (arrhythmias etc.). This suggests that patients are being sub-optimally unloaded and/or taking inadequate medical therapy and probably this decreases the chances for potential reverse remodeling and myocardial recovery. Moreover, a recent study demonstrated that cardiac dimensions obtained from echocardiography do not adequately reflect the degree of mechanical unloading of the heart. It has also shown strong evidence that pulmonary artery (PA) pressures monitoring can be reliably used to assess the pulmonary capillary wedge pressure (PCWP) and left ventricular end-diastolic pressure (LVEDP).

Symptomatic heart failure exacerbation requiring hospital admission may lie at the end of a spectrum of worsening hemodynamics that are unable to be detected before the manifestation of symptoms and limits the potential for myocardial recovery. Therefore, it is proposed that repeatedly adjusting LVAD pump flow speed and tailoring standard HF medications depending on the patient's PA pressure acquired from the CardioMEMS device can optimize pressure and volume unloading and promote reverse cardiac remodeling and recovery.

Clinical experience with LVAD support has shown that a subset of LVAD patients can experience reverse cardiac remodeling and significant improvement of myocardial function suggesting that LVAD-induced mechanical unloading of the failing heart may be a plausible therapeutic strategy aiming at myocardial recovery and device removal. These explanted patients have shown "myocardial plasticity" in clinical studies and that they can be responsive and sensitive to load changes. These patients will be carefully monitored to prevent increased load and wall stress to drive again the detrimental spiral of cardiac remodeling and HF recurrence, which appears to be the case in at least one third of LVAD patients after device weaning. Along the same lines, the results from another clinical study showed a significant and large reduction in hospitalization for HF patients who were managed with CardioMEMS. Therefore, further improvement of patients' HF management will depend mainly on better identification and pro-active management of their fluid and hemodynamic status. It is proposed that chronically adjusting HF medications using CardioMEMS-guided hemodynamic assessment in patients who have weaned from LVAD support could improve long-term durability of cardiac improvement after LVAD weaning.

ELIGIBILITY:
Inclusion Criteria:

* Severe clinical HF resistant to intensive medical therapy and requiring LVAD implantation
* Left ventricular ejection fraction <=25% and cardiomegaly at time of LVAD implantation
* Non-ischemic etiology of HF
* Undergone LVAD implantation within prior 4 weeks or planned for LVAD implant
* History of HF < 5 years
* Body Mass Index <=35 kg/m^2
* Pulmonary artery branch diameter between 7 - 15 mm
* Female subjects of childbearing age with negative urine or serum pregnancy test and agreeing to use reliable mechanical or hormonal form of contraception during study

Exclusion Criteria:

* Evidence of active acute myocarditis confirmed by histology
* History of previous cerebrovascular accident resulting in significant fixed motor deficit, limiting ability to perform exercise testing
* Implanted mechanical aortic and/or mitral valve(s) and/or right heart valve(s)
* Aortic valve closure
* Hypertrophic obstructive cardiomyopathy or sarcoidosis
* Left ventricular end-diastolic diameter below normal (restrictive cardiomyopathy)
* Irreversible multi-organ failure
* Diagnosis of psychiatric disease, irreversible cognitive dysfunction or poor psycho-social issues likely to impair compliance with study protocol
* Any condition that could limit survival to less than 2 years
* History of cardiac or other organ transplant
* Contraindicated to anti-coagulation, antiplatelet therapy, or diagnosis of coagulation disorders
* Require acute or chronic renal replacement therapy within 3 months prior to enrollment
* Participation in any other clinical investigations involving another Mechanical Circulating Support device or HF-related drug
* Active infection
* History of recurrent (>1) pulmonary embolism or deep vein thrombosis
* Unable to tolerate right heart catheterization
* Implantation of cardiac re-synchronization therapy < 3 months before enrollment
* Congenital heart disease
* Hypersensitivity or allergy to aspirin and/or clopidogrel

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2025-03-31 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects that meet explantation criteria by month 12 post-LVAD implantation, have LVAD explanted and retain left ventricular ejection fraction >=45% at 12 months post-LVAD weaning | 24 months
  Removal of LVAD happens when subject meets all five of the following explantation criteria: (1) left ventricular end-diastolic diameter < 60mm; (2) left ventricular end-systolic diameter < 50mm; (3) left ventricular ejection fraction > 45%; (4) left ventricular end-diastolic pressure <= 15 mmHg; (5) resting cardiac index > 2.4 L/min/m^2

SECONDARY OUTCOMES:
Hospital Admissions | 24 months
  Proportion of subjects admitted to the hospital for HF exacerbations at any time point during the study
Six-minute Walk Test | 12 months
  Subject performance during six-minute walk test at 12 months after LVAD implantation

CONTACTS AND LOCATIONS:
Overall Officials: Stavros Drakos, M.D., Principal Investigator — University of Utah
Locations (2):
- United States (2):
  - University of Kentucky, Lexington, Kentucky
  - Inova Heart and Vascular Institute, Falls Church, Virginia

IPD SHARING:
Plan to Share IPD: No